CLINICAL TRIAL: NCT06774846
Title: Aspirin in Acute Pneumonia in the Elderly: a Multicenter, Double-blind, Randomized, Placebo-controlled Trial.
Acronym: ASPAPY
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PUTOT PHRCN 2020
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Acute Pneumonia; Elderly Person
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Drug: Acetylsalicylic acid/Aspirin (100 mg)
- Control (Placebo Comparator)
  Interventions: Drug: Placebo acetylsalicylic acid (100 mg) / 0.9% sodium chloride

INTERVENTIONS:
Drug: Acetylsalicylic acid/Aspirin (100 mg) — Patients will receive 100 mg acetylsalicylic acid (or Aspirin) orally (tablet) once a day (or intravenously if oral administration is not possible in the acute phase of pneumonia), introduced within 84 hours of pneumonia diagnosis, for 90 days.
  Arms: Experimental
Drug: Placebo acetylsalicylic acid (100 mg) / 0.9% sodium chloride — patients in the placebo group will receive 100 mg placebo acetylsalicylic acid orally (tablet) once a day (or intravenously if oral administration is not possible in the acute phase of pneumonia), introduced within 84 hours of pneumonia diagnosis, for 90 days.
  Arms: Control

SUMMARY:
Acute pneumonia is a very common disease, and one of the leading causes of hospitalization and death in France. Almost a century after the discovery of penicillin, no major breakthrough has significantly reduced pneumonia-related mortality. While the choice of an appropriate antibiotic is decisive in the acute phase of the disease, the longer-term prognosis depends essentially on the worsening of other underlying pathologies, particularly in the elderly. In cured patients, excess mortality persists several months after the episode of pneumonia, due in particular to the onset of cardiovascular complications. Recent scientific literature shows an association between the prescription of cardio-protective drugs and survival after pneumonia. Older patients are usually excluded from interventional studies, so there are no specific recommendations for these patients at high risk of both acute pneumonia and cardiovascular events.

The aim of this study is to assess the efficacy of low-dose aspirin therapy after pneumonia in preventing cardiovascular events in the elderly.

The main objective is therefore to evaluate the impact of aspirin at a dose of 100mg per day on all-cause mortality at 90 days in patients over 75 years of age hospitalized for pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained from patient or relative/trusted person if patient unable to consent
* Age ≥75 years
* Clinical diagnosis of AP, presumed to be of bacterial or viral origin, with at least two of the following signs or symptoms:
* cough,
* purulent expectoration,
* thoracic pain,
* dyspnea/tachypnea,
* temperature > 37.8°C or < 36°C,
* unilateral crackles
* Patient hospitalized for at least 48 hours
* Onset of clinical signs < 7 days
* New radiological infiltrate documented by X-ray, ultrasound or CT scan

Exclusion Criteria:

* Mechanically ventilated pneumonia
* Documented SARS CoV2 pneumonia
* Patient with at least 3 episodes of inhalation pneumonitis in the 12 months prior to inclusion
* Pre-acute episode swallowing disorders impairing oral medication intake
* Physician-assessed life expectancy < 90 days
* Anticoagulant treatment (curative doses)
* Antiplatelet therapy
* Steroidal or non-steroidal anti-inflammatory treatment or oral corticosteroids without proton pump inhibitor (PPI)
* Treatment with methotrexate (>20 mg per week), anagrelide, probenecid, nicorandil, defibrotide
* Dyspepsia or gastroesophageal reflux disease (GERD) without PPI use
* Contraindications to aspirin (preventive doses) or its placebo at the time of inclusion:
* Hypersensitivity to acetylsalicylic acid or to any of the excipients of the investigational drug or placebo
* History of asthma induced by the administration of salicylates or non-steroidal anti-inflammatory drugs
* Active peptic ulcer disease or history of recurrent peptic ulcer disease
* History of cerebrovascular haemorrhage
* Previous gastrointestinal hemorrhage
* History of hemorrhage with Hemoglobin > 3g /dl requiring transfusion, vasoactive treatment or surgery
* Known hereditary or acquired coagulation disorder
* Thrombocytopenia (platelets < 50 giga/L)
* Acute kidney injury (clairance < 15 ml/min selon MDRD - Modification of Diet in Renal Disease),
* Liver cirrhosis or acute liver failure (PTT<50%),
* Severe uncontrolled heart failure
* Persistente severe hypertension (PAS > 180mmHg)
* Patient with mastocytosis
* Person not affiliated to a national social security scheme
* Patient under court protection

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 90 days after randomization